CLINICAL TRIAL: NCT02363712
Title: Biomechanical Therapy for Osteoarthritis of the Knee: a Randomized Controlled Trial(BIOTOK)
Brief Title: APOS Therapy for Osteoarthritis of the Knee: a Randomized Controlled Trial BIOTOK
Acronym: BIOTOK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Mäxi Foundation (Unknown); University of Bern (Other); Apos Medical and Sports Technology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 475_BIOTOK
Record Dates: First submitted 2015-01-29; First posted 2015-02-16 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, knee; therapy; shoe; Randomized Controlled Trial
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- APOS (Experimental): APOS(All Phase Of Step)-shoe
  Interventions: Device: APOS shoe
- Sham APOS (Sham Comparator): Sham APOS(All Phase Of Step)-shoe
  Interventions: Device: Sham-APOS shoe

INTERVENTIONS:
Device: APOS shoe — It consists of two shoes each with two large convex rubber balls called "Pertupods" screwed into the plantar surface of the sole so that a person walks on these balls.
  Arms: APOS
Device: Sham-APOS shoe — It has the same appearance as the APOS shoe, but without the rubber ball attachment on the plantar surface.
  Arms: Sham APOS

SUMMARY:
Painful knee osteoarthritis is common and treatments, short of knee replacement, are limited. The investigators plan to test the efficacy of a novel promising device for treatment of knee osteoarthritis affecting the inner part of the knee, the most common location. There are no disease modifying treatments available and therefore there is an emphasis on conservative management techniques to benefit individuals. Many of these treatments (insoles, braces, physiotherapy etc) have been shown to have relative success in individuals but a new novel device is demonstrating better effectiveness in this patient group. APOS (All Phases of Step) therapy consists of a shoe oriented system of care that works by shifting the load across parts of the knee and retraining the lower extremity muscles. Preliminary data suggest impressive favourable reductions in knee pain and a commensurate decrease in knee loading during walking. However, APOS treatment has never been evaluated in a randomised controlled trial even though it is widely used. The investigators propose to conduct a randomised blinded controlled trial of APOS treatment among persons with painful knee osteoarthritis affecting the inside (medial or lateral) of their knees. The investigators will focus on pain outcomes and quality of life. APOS has committed to provide the shoe system and a matched sham device, that they have developed, and will also provide the technicians trained to calibrate the pertupods (balls under the sole of the foot) on the shoe without charge. The research will be undertaken in a University setting for the gait evaluations.

DETAILED DESCRIPTION:
Background

Osteoarthritis (OA) is the most common arthritic condition and is one of the leading causes of disability in adults in Switzerland and worldwide (CDC 2009, WHO 2004). With the steady escalation of world life expectancy and constant decline in world birth rates, the incidence and prevalence of OA are expected to rise continuously worldwide throughout the years to come (Badley 1998). In Switzerland, OA is associated with decreased quality of life and frequent use of the health care system (Rosemann 2008).

Currently, no treatment can stop or reverse the progressive joint degeneration caused by OA. Most clinical interventions aim to improve pain and disability as these are the main symptoms afflicting OA patients (Grotle 2008), but managing pain associated with OA of the knee is difficult. Existing non-pharmacological and pharmacological interventions for OA remain insufficient. There are few effective nonsurgical treatments for painful knee OA (Jüni 2006).

OA affects different compartments in the knee, and biomechanical factors play an important role. Observational studies suggest that approximately 60% of affected persons have medial joint involvement (Niu 2009), which is subjected to excessive loading as quantified by the adduction moment across the knee. Bone marrow lesions (BMLs) are seen in knees in most persons with painful knee OA on fat suppressed MRI images. In the MOST cohort study, 80% of persons with medial knee OA and knee pain had medial BMLs. On histology, BMLs represent areas of bone damage with micro-cracks and remodelling. They are strongly related to malalignment such that knees with varus alignment have a high risk of BMLs in the medial compartment and those with valgus alignment have a risk of lateral BMLs (Felson 2003).

Wedges and orthotics which realign the knee have been tested in several randomized trials. This literature has undergone a Cochrane review of orthoses for treating knee OA (Brower 2005) which noted in its conclusion that, 'wearing a laterally wedged orthosis compared to wearing a neutral wedge may not lead to any difference in pain, knee function, or overall well-being'. None of the trials testing orthotics and inserts have shown any significant effect compared to control in terms of knee pain reduction. The other notable finding of almost all of these trials is that they reduced the varus moment across the knee, but by only 6% on average. One possible reason why inserts and orthotics have not worked to reduce pain is that they do not have a large enough realigning effect on the knee (as assessed by the varus moment).

APOS therapy, a new popular medical device, is a shoe system demonstrating potentially improved effectiveness in patients suffering from OA. This footwear has two potential mechanisms of action: 1. it can alter the pattern of knee loading, with reported reductions in the varus moment of 17% (Elbaz 2010), and 2. it retrains lower extremity motor control. Forcing people to avoid walking on the usual wide plantar surface and to instead walk on two rubber balls (APOS shoe) for half an hour at the start of the study, increasing successively (+10 min/week) up to almost 5 hours/day after 24 weeks (not exactly according to scheme but at the physiotherapist's discretion), forces muscular retraining and therefore serves as a built-in exercise intervention.

The investigators therefore aim to compare the efficacy and safety of APOS therapy in a large, pragmatic randomized controlled trial that includes gait analysis to understand the mechanistic action of the device.

Objective

Overall objective: The purpose of this trial is to evaluate whether APOS therapy can improve symptoms compared to Sham APOS therapy in participants with symptomatic knee OA.

Primary objective: The trial will determine the effect of APOS therapy on pain compared to Sham APOS therapy after 24 weeks.

Secondary objective: Secondary objectives will be to determine

* The effect of APOS therapy on pain compared to Sham APOS therapy after 4, 8, 12 and 16 weeks
* The effect of APOS therapy on joint stiffness, disability and overall assessment of the disease compared to Sham APOS therapy after 4, 8, 12, 16, and 24 weeks
* The effect of APOS therapy on quality of life after 4, 8, 12, 16, and 24 weeks
* The effect of APOS therapy on gait analysis measurements at baseline, after 4, 8, 12, 16 and 24 weeks
* The effect of APOS therapy on rescue analgesics compared to Sham APOS therapy throughout study duration (24 weeks) and after 24 weeks
* The time spent on average in the shoe

Methods

This trial is a patient-blind, single-centre, two-arm, parallel-group, 24 weeks (6 months) randomized controlled trial comparing APOS therapy and Sham APOS therapy. While the patients and physicians will be blinded regarding the intervention, the technician applying the shoes will not.

The trial will be conducted among persons with painful knee osteoarthritis. 220 patients will be randomly assigned on a 1:1 basis to one of the two treatments, APOS therapy or Sham APOS therapy. Randomisation will be stratified according to lateral / medial and unilateral / bilateral knee OA status.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant women
* Aged >= 40
* Outpatient setting
* ACR clinical criteria for OA of the knee
* Radiologically confirmed symptomatic uni- or bilateral OA of the knee for at least 6 months
* Radiological criteria: X-rays showing tibiofemoral knee osteoarthritis defined as at least Kellgren and Lawrence Grade 2
* At least moderate pain on the WOMAC pain scale (>3 on a standardized scale range from a minimum of 0 to a maximum of 10)
* Must understand German
* Informed Consent documented by participant signature

Exclusion Criteria

* Pregnant women
* Aged < 40
* History of an inflammatory rheumatic disease
* Non-knee musculoskeletal pain as or more severe than the knee pain
* Glucocorticoid injections in the knees in the previous three month
* Previous osteotomy
* Unilateral hemiprosthesis
* Unilateral total joint replacement
* Being treated for cancer
* Participation in another clinical trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
WOMAC pain subscale | End of treatment (at 24 weeks)

SECONDARY OUTCOMES:
WOMAC pain subscale | At week 4, 8, 12 and 16
WOMAC stiffness subscale | At baseline, at week 4, 8, 12, 16 and 24
WOMAC disability subscale | At baseline, at week 4, 8, 12, 16 and 24
Total WOMAC score | At baseline, at week 4, 8, 12, 16 and 24
Overall assessment of disease status on a 7 point likert scale | At baseline, at week 4, 8, 12, 16 and 24
  Data of this secondary outcome have never been collected.
Quality of life after using SF-36 | At baseline, at week 4, 8, 12, 16 and 24
Gait analysis | At baseline, at week 4, 8, 12, 16 and 24
  Consists of velocity, step length, single limb support and cadence
Self-reported health care utilisation | Up to 24 weeks
Rescue analgesics used | After 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Reichenbach, PD Dr. med., Principal Investigator — Institute of Social and Preventive Medicine (ISPM), University of Bern; Peter Jüni, Prof., Study Director — Applied Health Research Centre (AHRC), Li Ka Shing Knowledge Institute of St. Michael's Hospital, Department of Medicine and Institute of Health Policy, Management and Evaluation, University of Toronto, Canada
Locations (1):
- University of Berne, Bern, Switzerland

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence and most common causes of disability among adults--United States, 2005. MMWR Morb Mortal Wkly Rep. 2009 May 1;58(16):421-6. PMID 19407734
- [Background] Badley EM, Wang PP. Arthritis and the aging population: projections of arthritis prevalence in Canada 1991 to 2031. J Rheumatol. 1998 Jan;25(1):138-44. PMID 9458217
- [Background] Rosemann T, Grol R, Herman K, Wensing M, Szecsenyi J. Association between obesity, quality of life, physical activity and health service utilization in primary care patients with osteoarthritis. Int J Behav Nutr Phys Act. 2008 Jan 28;5:4. doi: 10.1186/1479-5868-5-4. PMID 18226211
- [Background] Grotle M, Hagen KB, Natvig B, Dahl FA, Kvien TK. Prevalence and burden of osteoarthritis: results from a population survey in Norway. J Rheumatol. 2008 Apr;35(4):677-84. Epub 2008 Feb 15. PMID 18278832
- [Background] Juni P, Reichenbach S, Dieppe P. Osteoarthritis: rational approach to treating the individual. Best Pract Res Clin Rheumatol. 2006 Aug;20(4):721-40. doi: 10.1016/j.berh.2006.05.002. PMID 16979535
- [Background] Niu J, Zhang YQ, Torner J, Nevitt M, Lewis CE, Aliabadi P, Sack B, Clancy M, Sharma L, Felson DT. Is obesity a risk factor for progressive radiographic knee osteoarthritis? Arthritis Rheum. 2009 Mar 15;61(3):329-35. doi: 10.1002/art.24337. PMID 19248122
- [Background] Felson DT, McLaughlin S, Goggins J, LaValley MP, Gale ME, Totterman S, Li W, Hill C, Gale D. Bone marrow edema and its relation to progression of knee osteoarthritis. Ann Intern Med. 2003 Sep 2;139(5 Pt 1):330-6. doi: 10.7326/0003-4819-139-5_part_1-200309020-00008. PMID 12965941
- [Background] Brouwer RW, Jakma TS, Verhagen AP, Verhaar JA, Bierma-Zeinstra SM. Braces and orthoses for treating osteoarthritis of the knee. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD004020. doi: 10.1002/14651858.CD004020.pub2. PMID 15674927
- [Background] Elbaz A, Mor A, Segal G, Debbi E, Haim A, Halperin N, Debi R. APOS therapy improves clinical measurements and gait in patients with knee osteoarthritis. Clin Biomech (Bristol). 2010 Nov;25(9):920-5. doi: 10.1016/j.clinbiomech.2010.06.017. Epub 2010 Jul 16. PMID 20637534
- [Background] Bar-Ziv Y, Beer Y, Ran Y, Benedict S, Halperin N. A treatment applying a biomechanical device to the feet of patients with knee osteoarthritis results in reduced pain and improved function: a prospective controlled study. BMC Musculoskelet Disord. 2010 Aug 10;11:179. doi: 10.1186/1471-2474-11-179. PMID 20698991
- [Background] Trelle S, Reichenbach S, Wandel S, Hildebrand P, Tschannen B, Villiger PM, Egger M, Juni P. Cardiovascular safety of non-steroidal anti-inflammatory drugs: network meta-analysis. BMJ. 2011 Jan 11;342:c7086. doi: 10.1136/bmj.c7086. PMID 21224324
- [Derived] Reichenbach S, Felson DT, Hincapie CA, Heldner S, Butikofer L, Lenz A, da Costa BR, Bonel HM, Jones RK, Hawker GA, Juni P. Effect of Biomechanical Footwear on Knee Pain in People With Knee Osteoarthritis: The BIOTOK Randomized Clinical Trial. JAMA. 2020 May 12;323(18):1802-1812. doi: 10.1001/jama.2020.3565. PMID 32396180